CLINICAL TRIAL: NCT04664686
Title: Rate or Rhythm Control in CRT: the RHYTHMIC Study
Acronym: RHYTHMIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 265388
Record Dates: First submitted 2020-12-10; First posted 2020-12-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AF catheter ablation (Active Comparator)
  Interventions: Procedure: AF catheter ablation
- AV node ablation (Active Comparator)
  Interventions: Procedure: AV node ablation

INTERVENTIONS:
Procedure: AF catheter ablation — Isolation of all four pulmonary veins and additional lesions, considered indicated by the operator
  Arms: AF catheter ablation
Procedure: AV node ablation — AV node ablation
  Arms: AV node ablation

SUMMARY:
70 patients with heart failure, AF and CRT with BiV<95% will be randomised to either AF ablation or AV node ablation. Evaluation at 6 months with echocardiography and clinical assessment.

DETAILED DESCRIPTION:
70 patients with heart failure, AF and CRT with BiV<95% will be recruited from outpatient clinic, pacing clinic or inpatient wards. Patients will be consented and will undergo baseline investigation with a transthoracic 2D echocardiogram, ECG, blood tests, cardiac CT with perfusion imaging, 6 minute walk test (6MWT), cardio-pulmonary exercise test (CPET) and Minnesota Living with Heart Failure Questionnaire. Patients who are successfully screened will be randomized 1:1 to receive AF catheter ablation rhythm control or AV-node ablation rate control.

Ablation Procedure:

Patients will receive either AF catheter ablation or AV-node ablation during the procedure. Patients randomised to AF catheter ablation will receive isolation of all four pulmonary veins and additional lesions, considered indicated by the operator. The procedure will be classified as successful if all four veins are isolated and the patient is in sinus rhythm. Patients may undergo DC-cardioversion under sedation if they remain in atrial fibrillation. AV-node ablation will be performed in line with current standard of care. Patients will also undergo additional research investigations at the time of ablation as follows:

Acute Haemodynamic Study:

All patients will also undergo an acute haemodynamic study with pressure wire assessment of both the right ventricle and the left ventricle at the start and end of the procedure. This involves inserting pressure wires into the RV via a vein in the groin and into the LV via an artery in the wrist or the groin. This will provide novel information on how AF catheter ablation and AV-node ablation affect cardiac contractility.

Invasive Electroanatomical Mapping (Optional):

This is an optional additional procedure that patients may opt into at the time of recruitment. This is performed during the ablation procedure with mapping catheters and software which are CE marked and already in clinical use. Mapping of all four cardiac chambers will be performed. This will be achieved via a vein and an artery in the groin. This will provide novel information on how AF catheter ablation and AV-node ablation affect electrical activation of the atria and ventricles.

Follow-up:

Patients will undergo a 2D transthoracic echocardiogram and ECG 1 week post ablation. Patients will then be followed up at 6 months with 2D transthoracic echocardiogram, ECG, clinical review, CPET, 6MWT, Minnesota Living with Heart Failure Questionnaire and pacing check.

Patients in the AF catheter ablation group who have a recurrence of AF after a 3 month blanking period will be permitted a re-do procedure. The follow-up investigations will take place 6 months after the re-do procedure. If a patient has recurrence of AF after a second ablation procedure and it is felt a third procedure is indicated, this will be performed after the six month follow-up period has ended and the patient is no longer in the study. They will be included in the intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent to participate and willing to comply with the clinical investigation plan and follow-up schedule.
* QRS duration >120ms on surface ECG, severe left ventricular systolic impairment (EF≤35%) and clinical symptoms of heart failure despite optimum medical therapy (NYHA class II-IV) at time of CRT implant or upgrade
* Successful CRT implant or upgrade including atrial lead
* Biventricular pacing percentage <95% secondary to atrial fibrillation at least 3 months post implant or upgrade
* Clinically indicated for AV node ablation

Exclusion Criteria:

* Life expectancy <1 year
* Presence of atrial or ventricular thrombus
* Permanent atrial fibrillation
* Mechanical aortic valve replacement
* Severe peripheral vascular disease
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
* Participation in other studies with active treatment / investigational arm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Difference in ejection fraction | 6 months
  On 2D echocardiography

SECONDARY OUTCOMES:
Difference in left ventricular end systolic volume | 6 months
  On 2D echocardiography
Difference in biventricular pacing percentage | 6 months
  On pacemaker check
Difference in quality of life | 6 months
  Assessed by Packer's Clinical Composite Score
Difference in NYHA class | 6 months
  On clinical assessment
Difference in heart failure symptoms | 6 months
  Assessed by Minnesota Living with Heart Failure Questionnaire
Difference in 6-minute walk test | 6 months
Difference in VO2 max | 6 months
  Assessed via cardio pulmonary exercise test (CPET)
Difference in AF burden | 6 months
  Assessed via pacing check

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Rinaldi, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas' NHS Foundation Trust, London, United Kingdom